CLINICAL TRIAL: NCT05048693
Title: Use of New Antibiotics Against Multidrug-resistant Gram-negative Bacteria in Swedish University Hospitals
Brief Title: Use of New Antibiotics in Sweden
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Karolinska University Hospital (Other); Sahlgrenska University Hospital (Other); University Hospital, Linkoeping (Other); Skane University Hospital (Other); University Hospital, Umeå (Other); Örebro University, Sweden (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01678
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Multi-antibiotic Resistance
Keywords: Multidrug-resistant Gram-negative bacteria; Antibiotic resistance; Cefiderocol; Ceftazidime-avibactam; Ceftolozane-tazobactam; Fosfomycin; Meropenem-vaborbactam; Imipenem-relebactam

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Antibiotic resistance is a growing global health problem of great concern, especially multidrug-resistant Gram-negative bacteria. In recent years some new antibiotics targeting these bacteria have been developed. The aim of this study is to investigate how these new antibiotics are used in Sweden. Information will be collected on patients, types of infections, dosing strategies, treatment outcome and occurrence of antibiotic resistance during treatment. The overall goal is to increase the knowledge about how these antibiotics are prescribed and how to optimize the use of them in clinical practice.

DETAILED DESCRIPTION:
Emergence and spread of antibiotic-resistant bacteria is one of the greatest threats facing human health today. Multi-resistant Gram-negative bacteria constitutes the biggest challenges and particularly carbapenem-resistant bacteria, against which available treatment options usually are very limited and the mortality is high (>50%) in severly ill patients. In recent years some new antibiotics have been developed with in-vitro effect against those bacteria. Still, clinical data regarding those antibiotics are limited and resistance development has been reported. Combination therapy with two or more antibiotics are often used to treat multi-resistant Gram-negative bacteria and are sometimes applied also with the newer drugs. Combination therapy is supported mainly by in vitro studies rather than clinical evidence. More research is needed to investigate which antibiotic combinations has the biggest potential.

The main objective of this study is to assess current use of the following antibiotics in Swedish university hospitals: cefiderocol, ceftazidime-avibactam, ceftolozane-tazobactam, fosfomycin, meropenem-vaborbactam and imipenem-relebactam.

Following informed consent, all patients treated with any of the study drugs at one of the seven university hospitals in Sweden can be included in the study. Guardian approval is needed to include study participants <15 years of age. Besides routine testing with biomarkers and cultures within clinical practice, bacterial cultures will be taken seven days after start of treatment with the study drug, from the sample site where the infecting pathogen was first identified (e.g., blood, wound, nasopharynx, urine), to assess microbiological cure. Screening for multidrug-resistant Gram-negative bacteria in feces will also be conducted with screening cultures seven days after initiated therapy with study drug to detect emergence of resistance in the intestinal microbiota. The cultures will be analyzed at the local clinical microbiology departments.

Information on patient characteristics (age, gender, comorbidity etc.), site of infection, infecting pathogen and associated resistance profile, severity of infection, choice of treatment (drug, dose, treatment duration and eventual antibiotic combination therapy) will be obtained from the electronical medical records. Further treatment outcome including mortality, treatment failure, increasing need of intensive care, duration of hospitalization, suspected side effects and occurrence of Clostridioides difficile enteritis will also be extracted. The follow-up period is 30 days.

Patient names and personal identification numbers will be replaced by a number. Personal data will be stored at the Department of infectious diseases, at respective hospital where the study participant has been included. Only the responsible researchers will have access to the code key and be able to link personal information to the individual participants. All information will be handled in accordance with the General Data Protection Regulation (GDPR) and all analyses and presentation of data will be performed using anonymous data.

To determine antibiotic resistance profiles of the infecting pathogens, bacterial isolates will be sent to the reference laboratory at Uppsala University. The strains will be characterized with phenotypical methods for minimum inhibitory concentration (MIC) determination (e.g., microdilution, agar dilution) as well as genetical testing with whole-genome sequencing determining the presence of resistance genes and genetic mutations (e.g., production of beta lactamases, porin loss and efflux). In case of repeated growth of the same bacterial species in clinical or screening samples seven days from start of treatment, the two strains (prior and post treatment start of study drug) will be compared by MIC determination and whole-genome sequencing to detect emergence of antibiotic resistance during treatment.

Finally, the isolates will undergo in-vitro testing at the reference laboratory at Uppsala University, where the efficacy of different antibiotic combinations will be investigated with multiple in vitro methods including automated time-lapse microscopy and bacterial time-kill experiments with static and dynamic antibiotic concentrations. Bacterial killing, bacterial growth and selection of resistant subpopulations will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with any of the following antibiotics; cefiderocol, ceftazidim-avibactam, ceftolozan-tazobactam, fosfomycin, meropenem-vaborbactam or imipepenem-relebactam against an acute infection.

Exclusion Criteria:

* Ongoing treatment with any of the above mentioned antibiotics for more than seven days at the point of inclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in seven University Hospitals in Sweden treated with any of the following antibiotics; cefiderocol, ceftazidim-avibactam, ceftolozan-tazobactam, fosfomycin, meropenem-vaborbactam or imipepenem-relebactam against an acute infection.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Clinical cure | 30 days from enrollment
  Defined as discontinuation of the study drug following clinical or laboratory improvement with regard to the treated infection. Information on this will be extracted from the electronical medical records.
Microbiological cure | 30 days from enrollment
  Defined as negative follow-up clinical cultures sampled seven days from start of treatment with the study drug. Information on this will be extracted from the electronical medical records.
All-cause mortality | 30 days from enrollment
  Defined as death within 30 days from start of treatment with the study drug. Information on this will be extracted from the electronical medical records.

SECONDARY OUTCOMES:
Severity of illness | 30 days from enrollment
  The severity of illness will be assessed with Sequential Organ Failure Assessment (SOFA) Score, which is a scoring system used in the assessment of acute morbidity in a range of critical illnesses. The SOFA-score allows for calculation of both the number and the severity of organ dysfunction in six organ systems (respiratory, coagulation, liver, cardiovascular, renal, and neurologic) and assigns a score based on the data obtained in each category. The higher the SOFA score, the higher the likely mortality. The requested information to calculate the score for each participant will be obtained from the electronical medical records.
Indication for treatment | 30 days from enrollment
  The type of infection will be obtained from the electronical medical records. The clinical assessment of infection type will be based on clinical symptoms and the sample site of cultures where the infecting bacteria was identified (e.g., blood, wound, nasopharynx, urine).
Use of antibiotic combination therapy | 30 days from enrollment
  Information on any concomitant antibiotic treatment used in combination with the study drug will be obtained from the electronical medical records.
Microbiological results | 30 days from enrollment
  Results from routine microbiological analyses (bacterial species, antibiotic susceptibility) of infecting bacteria will be obtained from the electronical medical records.
Treatment failure | 30 days from enrollment
  Defined as change of antibiotic treatment against infecting bacteria because of treatment failure with the study drug as documented by the treating physician. Information on this will be extracted from the electronical medical records.
Colonization with multidrug-resistant Gram-negative bacteria in feces | 30 days from enrollment
  Screening of multidrug-resistant Gram-negative bacteria in fecal samples will be performed seven days after start of treatment with the study drug to detect emergence of antibiotic resistance in the intestinal microbiota. Information on screening results will be obtained from the electronical medical records.
Mortality attributable to infection | 30 days from enrollment
  Defined as death within 30 days from start of treatment with the study drug where the cause of mortality is determined to be the infection treated with the study drug, as documented by the treating physician. Information on this will be extracted from the electronical medical records.
Readmissions within 30 days | 30 days from enrollment
  Information on readmissions within 30 days from start of treatment with the study drug will be obtained from the electronical medical records.
Documented side effects | 30 days from enrollment
  Information on suspected side effects associated with treatment with the study drug will be obtained from the electronical medical records.
Occurrence of Clostridioides difficile infection | 30 days from enrollment
  Information on confirmed Clostridioides difficile infection within 30 days from start of treatment with the study drug will be obtained from the electronical medical records.
Duration of hospitalization | 1 year from enrollment
  Information on number of hospital days will be obtained from the electronical medical records.
Use of study drug in relation to the approved indications | 1 year from enrollment
  Indication for the prescribed study drug (secondary outcome measure no. 2) will be compared to the approved indications for the respective study drug according to the summary of product characteristics (SPC).
Dosing of study drug in relation to recommendations | 1 year from enrollment
  Dosing of the study drug, extracted from the electronical medical records, will be compared to the approved dosing according to the summary of product characteristics (SPC).
Phenotypic characterization of isolated bacteria | 1 year from enrollment
  Isolated bacteria will be collected from the local microbiological laboratories for minimum inhibitory concentration (MIC) determination with phenotypical methods (e.g., microdilution, agar dilution) at the reference laboratory at Uppsala University.
Genotypic characterization of isolated bacteria | 1 year from enrollment
  Isolated bacteria will be collected from the local microbiological laboratories for genotypic characterization by whole-genome sequencing to determine the presence of resistance genes and mutations (e.g., production of beta-lactamases, porin loss and efflux) at the reference laboratory at Uppsala University.
Emergence of antibiotic resistance | 2 years from enrollment
  In case of repeated growth of the same bacterial species in clinical or screening samples seven days from start of treatment, the two isolates (prior and post treatment start with study drug) will be compared by MIC determination and whole-genome sequencing at the reference laboratory at Uppsala University regarding resistance genes and mutations to detect resistance development during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Tängdén, MD, Phd, Principal Investigator — Uppsala University Hospital
Locations (7):
- Sweden (7):
  - Sahlgrenska University Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Lund
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, Stockholm
  - Umeå University Hospital, Umeå
  - Uppsala University Hospital, Uppsala